CLINICAL TRIAL: NCT06354738
Title: Improving Endometrial Cancer Assessment by Combining the New techniqUe of GENomic Profiling With Surgical Extra uterIne disEase Assessment
Brief Title: Improving Endometrial Cancer Assessment by Combining Genomic Profiling and Surgical Assessment
Acronym: EUGENIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Frederic Amant, Head of the scientific Unit of Gynecologic Oncology, Full professor at Faculty of Medicine and Clinical Staff Specialist at Gynecological Oncology at UZ Leuven, Full professor at Faculty of Medicine, University of Amsterdam, University Hospital, Gasthuisberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S66928
Record Dates: First submitted 2024-03-21; First posted 2024-04-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Genomic profiling; Molecular classification; Disease staging
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All women older than 18 newly diagnosed with endometrial cancer of all stages and histotypes (Experimental): All patients must undergo total hysterectomy and bilateral salpingo-oophorectomy or bilateral salpingectomy if premenopausal status and the lymph-node assessment according to European guidelines and local protocol. A comprehensive surgical peritoneal staging is required, which includes omentectomy/omental biopsies and six peritoneal biopsies.
  Interventions: Procedure: total hysterectomy with bilateral salpingo-oophorectomy, lymph node staging and comprehensive peritoneal staging

INTERVENTIONS:
Procedure: total hysterectomy with bilateral salpingo-oophorectomy, lymph node staging and comprehensive peritoneal staging — Surgical treatment will consist of total hysterectomy with bilateral salpingo-oophorectomy according to international guidelines.
  In low- and intermediate-risk EC patients, staging will include a sentinel lymph node (SLN) procedure. In high intermediate-risk and high-risk EC patients, lymph node staging will involve SLN procedure and/or pelvic and para-aortic lymph node dissection (LND), depending on the local protocol.
  The Study-related procedures include infracolic omentectomy or two separate omental representative biopsies, biopsies of all suspicious lesions as well as six peritoneal sites (bladder, pouch of Douglas, bilateral paracolic gutter and bilateral diaphragm).
  Stage IV patients will be treated according to European guidelines. When feasible, full surgical intervention (i.e. debulking) is recommended. If this cannot be achieved, a radiologic and/or histologic confirmation of tumor spread beyond the uterus will be accepted.

SUMMARY:
EUGENIE is a prospective multicentre interventional study, focused on improving endometrial cancer (EC) assessment by combining the new technique of genomic profiling with surgical extra uterine disease assessment. The investigators aim to correlate EC stage to each of the molecular subgroups of disease and thereby guide surgical treatment and staging of EC by determining the association between molecular classification and disease stage and evaluating if and how disease stage in each of the molecular subgroups associates with prognosis.

DETAILED DESCRIPTION:
Current treatment for endometrial cancer (EC) includes a hysterectomy with bilateral salpingo-oophorectomy. Further surgical staging procedures (lymphadenectomy, peritoneum, and/or omentum biopsies) can be performed in order to detect metastases and determine the disease stage. The type and extent of this surgical staging depend on a pre-operative risk assessment and guides adjuvant treatment (chemo- or radiotherapy). However, this pre-operative risk assessment based on histology and imaging is relatively inaccurate: first, preoperative histology presents high intersubjective variability leading to poor reproducibility in the assignment of histotype and the concordance between preoperative histology and final histology is poor. In addition, preoperative imaging modalities are expensive, time-consuming, hampered by non-perfect accuracies, require specialized expertise, or present limitations in reproducibility and availability. As a result, this leads to an incorrect risk estimation of metastases at diagnosis in EC patients with a consequent over- or undertreatment of patients. Thus, there is an urgent need to develop risk stratification strategies that will better predict the presence and localization of metastases in EC patients and therefore more efficiently tailor surgical staging procedures.

In 2013 The Cancer Genome Atlas (TCGA) Research Network developed a new molecularly driven classification system, that divides EC tumours into the well-known four molecular subgroups (POLE, MMRd, p53abn, NSMP) and has shown to surpass histologic subtyping and grading to more efficiently predict prognosis. However, the relation between the four molecular subgroups and the risk of tumour spread beyond the uterus at diagnosis has insufficiently been investigated so far and, as a consequence, surgical staging should not yet be adapted based on the molecular endometrial cancer subtype.

Thus, new studies are needed to assess the value of surgical staging in this molecular era and EUGENIE Study has been developed to bridge this knowledge gap.

The investigators believe that the future is in integrating morphologic and molecular findings, so the preoperative diagnosis will also support accurate surgical decision making and therefore a more tailored management of all EC patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained before any screening procedures
* Women ≥ 18 years
* First diagnosis of EC, all disease stages and all histo-types

Exclusion Criteria:

* Participant has a history of pelvic or para-aortic lymph node dissection or sampling, previous pelvic (and/or para-aortic) radiotherapy, previous neoadjuvant chemotherapy
* Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
* Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Endometrial cancer stage | 72 months
  Endometrial cancer stage assessed according to the 2009 an 2023 International Federation of Gynecology and Obstetrics (FIGO) staging
Molecular type of endometrial cancer | 72 months
  Tumor classification using the molecular classification as proposed by either ProMisE or TRANSPORTEC.
  Groups will be classified as follows:
  1. MMR: Mismatch Repair Protein Status will be determined as a surrogate for microsatellite instability (MSI) by considering the immunohistochemical (IHC) staining of the MMR proteins. In case of loss of staining of one or more MMR proteins, the EC will be classified as MMR deficient (MMRd), otherwise, the carcinoma will be coded as MMR proficient (MMRp).
  2. POLE: if the POLE exonuclease domain mutations (EDM) gene is mutated (i.e. a pathogenic mutation), the tumour will be classified as POLE.
  3. p53 IHC: TP53 mutation status will be determined via IHC and in case of inconclusive p53 staining, also sequencing.
  4. NSMP: a carcinoma that has not been stratified into groups 1), 2) or 3) will be categorized into the NSMP (no specific molecular profile or copy number low).

SECONDARY OUTCOMES:
Overall survival | 72 months
  Overall survival
Time to recurrence | 72 months
  Time to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Amant, MD, PhD, Principal Investigator — UZ Leuven Gasthuisberg
Locations (1):
- UZ Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Protocol — https://pubmed.ncbi.nlm.nih.gov/36977506/